CLINICAL TRIAL: NCT01990456
Title: Strategies for Optimal Lung Ventilation in ECMO for ARDS: The SOLVE ARDS Study
Acronym: SOLVE ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Eddy Fan, MD, PhD, University of Toronto
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SOLVE ARDS_01
Record Dates: First submitted 2013-11-06; First posted 2013-11-21 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Extracorporeal Membrane Oxygenation; Ventilator-Induced Lung Injury; Ventilators, Mechanical; Pulmonary Heart Disease; Ultrasonography
MeSH Terms: conditions — Respiratory Distress Syndrome; Ventilator-Induced Lung Injury; Pulmonary Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PHASE 1: impact of tidal ventilation on VILI (Experimental): In the first phase we will test whether administering a distending inspiratory pressure to produce tidal ventilation is superior to a strategy where only continuous positive airway pressure (CPAP) is applied for ventilation induced lung injury (VILI) mitigation, as assessed by its impact on biotrauma (serum cytokines) and physiologic measurements.
  Interventions: Device: PHASE 1: impact of tidal ventilation on VILI
- PHASE 2: impact of PEEP on VILI (Experimental): In the second phase we will gain more insight as to whether a strategy that utilizes a PEEP level that correspond to best compliance is beneficial over Zero End-Expiratory Pressure (ZEEP). We will test the impact of both strategies on biotrauma (serum cytokines), physiologic parameters, and right ventricular function (transesophageal echocardiographic assessment).
  Interventions: Device: PHASE 2: impact of PEEP on VILI

INTERVENTIONS:
Device: PHASE 1: impact of tidal ventilation on VILI — PHASE 1A - Baseline - Standard Ventilation Protocol (PCV 10 cmH2O, PEEP 10 cmH2O, RR 10, FiO2 0.30) PHASE 1B - CPAP Strategy - CPAP 10 cmH2O for 1 hour PHASE 1C - Higher Tidal Ventilation Strategy (PCV 20 cmH2O, PEEP 10 cmH2O, RR 10, FiO2 0.30) PHASE 1D - Return to Baseline - Standard Ventilation Protocol
  Arms: PHASE 1: impact of tidal ventilation on VILI
Device: PHASE 2: impact of PEEP on VILI — PHASE 2A - Baseline - Standard Ventilation Protocol - (PCV 10 cmH2O, PEEP 10 cmH2O, RR 10, FiO2 0.30) PHASE 2B - Decremental PEEP Trial PHASE 2C - CPAP set at best compliance of respiratory system (as per decremental PEEP Trial) PHASE 2D - ZEEP PHASE 2E - Return to Baseline - Standard Ventilation Protocol
  Arms: PHASE 2: impact of PEEP on VILI

SUMMARY:
Due to lack of studies on mechanical ventilation strategies in patients with severe Acute Respiratory Distress Syndrome (ARDS) supported with Veno-Venous Extra-Corporeal Membrane Oxygenation (VV ECMO), ventilator settings in this patient population are set arbitrarily.

In this two-phases prospective, interventional, pilot study we hope to gain physiologically relevant data on two aspects of mechanical ventilation in patients with severe ARDS supported with VV ECMO: (1) the use of tidal ventilation and (2) the level of Positive End-Expiratory Pressure (PEEP).

1. PHASE 1: impact of tidal ventilation on VILI (10 patients) We hypothesized that a CPAP strategy that minimizes end-tidal pulmonary stress and strain mitigates VILI compared to the current mechanical ventilation practice that employs tidal ventilation in patients with severe ARDS on ECMO.

   In this first phase we will test whether administering a distending inspiratory pressure to produce tidal ventilation is superior to a strategy where only continuous positive airway pressure (CPAP) is applied for ventilation induced lung injury (VILI) mitigation, as assessed by its impact on biotrauma (serum cytokines) and physiologic measurements.
2. PHASE 2: impact of PEEP on VILI (10 patients) We also hypothesized that adjusting PEEP to maximize respiratory system compliance reduces VILI in patients with severe ARDS on ECMO.

In the second phase we will therefore gain more insight as to whether a strategy that utilizes a PEEP level that correspond to best compliance is beneficial over Zero End-Expiratory Pressure (ZEEP). We will test the impact of both strategies on biotrauma (serum cytokines), physiologic parameters, and right ventricular function (transesophageal echocardiographic assessment).

Because ARDS patients supported with VV ECMO can be hemodynamically unstable, the use of imaging techniques that require transport, such as computed tomography, is limited. Therefore, bedside imaging techniques, such as pleural and lung ultrasound (PLUS) and focused bedside cardiac ultrasonography, are important tools for clinicians who care for these patients. This study will allow us to learn whether these techniques are feasible and valid in this patient population.

Furthermore, the knowledge gained from this study will allow us to assess the rationale and feasibility of performing a similar larger, randomized study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Severe ARDS (Berlin Definition)
* VV ECMO < 72 hours
* Endotracheal intubation or tracheostomy

Exclusion Criteria:

* Thoracic surgery/lung transplantation during the current hospitalization
* Contraindications to a RM (MAP < 60 mmHg despite administration of fluids and vasopressors; Active air leak through a thoracostomy tube; Pneumothorax, or subcutaneous or mediastinal emphysema, (if chest tube has not been inserted))
* Contraindications to TEE
* Age < 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Induced Lung Injury (VILI) in patients with ARDS on ECMO ventilated with different strategies (tidal ventilation, CPAP, ZEEP), as measured by Serum Cytokines | 1 hour after initiation of each experimental ventilation strategy

SECONDARY OUTCOMES:
Impact of a CPAP strategy (PEEP set at best compliance and at ZEEP) in patients with severe ARDS on ECMO, as measured by transesophageal echocardiography (TEE) | 30 minutes after initiation of experimental CPAP/ZEEP strategy
  Quantification of RV function:
  1. RVEDA/LVEDA
  2. LV end-diastolic/systolic eccentricity indexes:
  3. 2D RVFAC
  4. TAPSE
  5. Tissue Doppler-derived tricuspid lateral annular systolic velocity (S')
  6. RIMP
  7. 3D EF < 44%
  8. Myocardial Acceleration During Isovolumic Contraction
  9. Regional RV Strain
Feasibility and validity of focused cardiac ultrasound, as compared to TEE as gold standard, in the assessment of RV function in patients with ARDS on ECMO | 30 minutes after initiation of experimental CPAP/ZEEP strategy
  Quantification of RV function:
  1. RVEDA/LVEDA
  2. TAPSE
  3. RV Annular Velocity (S')
  4. LV end-diastolic and end-systolic eccentricity indexes
Feasibility of lung ultrasound in patients with severe ARDS on ECMO | 30 minutes after initiation of experimental CPAP/ZEEP strategy
  Lung Ultrasound Score
Feasibility (patient recruitment, protocol adherence, physiologic tolerability) | At overall study completion (i.e., 24 months from study start or after enrolment of last patient)
  This outcome will be assessed by:
  * the ability to enrol the proposed patient sample within the timeframe of the study (24 months)
  * >90% adherence to the experimental protocol on enrolled patients
  * >80% completion of the entire experimental protocol on enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fan, MD, PhD, Principal Investigator — University Health Network, University of Toronto; Niall D. Ferguson, MD, MSc, Principal Investigator — University Health Network, University of Toronto
Locations (1):
- Medical Surgical ICU - Toronto General Hospital, Toronto, Ontario, Canada